CLINICAL TRIAL: NCT04460690
Title: Rapid, Onsite COVID-19 Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); AIDS Vaccine Research Lab (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0855; A536300 (Other: UW Madison); SMPH/PATHOL-LAB MED/ANAT PATH (Other: UW Madison); Protocol Version 8/30/2020 (Other: UW Madison); 5P51OD011106-59 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-07-07 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Sars-CoV2
Keywords: rapid detection; assay; saliva; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Rapid Onsite COVID-29 Testing (Experimental): Community participants provide a saliva sample for a simple test to detect high concentrations of SARS-CoV-2 in saliva with assays that require no specialized equipment and can be completed in one hour.
  Interventions: Device: Rapid Onsite COVID-19 Detection

INTERVENTIONS:
Device: Rapid Onsite COVID-19 Detection — saliva assay test for high concentrations of SARS-CoV-2

SUMMARY:
The purpose of this research study is to evaluate and improve a rapid COVID-19 test. The test is designed to identify people who are most contagious and likely to spread the virus to others. This test will be performed at various locations in the Madison area using a mobile laboratory or standard lab space for processing. Saliva samples can be collected and processed at these locations or participants can self-collect at home and drop their samples off at designated locations for same day processing. Results of potential findings of clinical significance will be communicated to the participants by a physician with appropriate expertise on the study team. Individuals with a potential finding of clinical significance will be encouraged to self-isolate and obtain a diagnostic test at their earliest convenience. No results will be given if the test is negative. If the participant consents, advanced molecular testing such as PCR or viral sequencing can be done and results can be shared via online databases, presentations and publications along with the date, site and county of collection to help facilitate tracking the spread of the virus.

DETAILED DESCRIPTION:
Virtually all COVID-19 RNA assays require centralized laboratories. Samples collected in locations including public testing sites, workplaces, nursing homes, and residential housing are transported to centralized laboratories for testing, leading to lengthy delays in results reporting. The window of maximal contagiousness is thought to be only a few days, so these delays create the risk of excess transmission. Current testing methods are painful, which encourages testing hesitancy. Rapid, onsite detection of SARS-CoV-2 RNA from non-invasive saliva could overcome these issues and provide a pathway to high-throughput detection of people at the greatest risk of SARS-CoV-2 transmission but the logistics of such a testing program require real-world prototyping.

The investigators have developed a simple test to detect high concentrations of SARS-CoV-2 in saliva with assays that require no specialized equipment and can be completed in one hour. This assay is not diagnostic for SARS-CoV-2; instead, it specifically identifies saliva samples that have high amounts of viral RNA that are correlated with live virus shedding. Many samples that would be identified as SARS-CoV-2 by diagnostic qRT-PCR would be negative with this saliva assay. Conversely, detection of RNA in saliva is a potential finding of clinical significance, so participants with that result will be contacted by a medical professional to discuss potential follow-up with their own health care provider, including a possible independent diagnostic testing.

Because the assay requires no specialized equipment, it can be performed at the site of sample collection using a portable laboratory that fits in the backseat of a car. The prototype testing will take place in a variety of settings that may include parking lots, workplaces, nursing homes and residential housing. Participants will be asked to consent to provide a saliva sample that will be tested for SARS-CoV-2 RNA levels consistent with live virus shedding. The consent document will explicitly state that this is not a diagnostic test for SARS-CoV-2 but that a potential finding of clinical significance should be discussed with a medical professional. Participants can opt-out of receiving any results at the time of consent and can provide samples for the sole purpose of contributing to community surveillance and assay development. Paper consent forms will be reviewed and signed and held by team members in a secure location (locked box at the collection site) until taken back to the AIDS Vaccine Research Laboratory for storage. Participants will then spit into a coded vessel (e.g., cup or tube). Samples should be at least 1ml (~¼ teaspoon) and will be assayed for the presence of SARS-CoV-2 RNA using the aforementioned detection assay; the presence of high concentrations of SARS-CoV-2 RNA is indicated by a colorimetric change from pink to yellow/orange.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Willing to provide informed consent and spit into a vessel
* Individuals at least 5 years of age and have a parent or legal guardian present to consent if under 18 years
* Adult participants must have decision-making capacity to provide consent on their own behalf.
* Participants must be able to speak English

Exclusion Criteria:

* Under 18 years of age with no parent or legal guardian present or under the age of 5 yrs
* Participants must not have visual or hearing impairments, or low literacy, that would prevent them from reading the consent form and interacting with a member of the research team to ask questions and receive responses during the consent process

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O'Connor, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will consent to having their data (not their name) and viral sequences shared with the public via manuscripts, presentations and online databases; the study team will share that with other researchers when needed. Samples can be shared with UW researchers internally and non UW researchers through the Material Transfer Agreement process.
Time Frame: Data from this study may be requested from other researchers 7 years after the completion of the primary endpoint by contacting David O'Connor at the University of Wisconsin - Madison.

REFERENCES:
- See also: Dave O'Connor's Lab — https://dho.pathology.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapid Onsite COVID-29 Testing
Started | 93
Community Participants | 83
Investigator Participants | 10
Completed | 93
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Rapid Onsite COVID-29 Testing - Investigators; Rapid Onsite COVID-29 Testing - Participants: Community participants provide a saliva sample for a simple test to detect high concentrations of SARS-CoV-2 in saliva with assays that require no specialized equipment and can be completed in one hour.
  Rapid Onsite COVID-19 Detection: saliva assay test for high concentrations of SARS-CoV-2
- Total: Total of all reporting groups
Arm/Group | Rapid Onsite COVID-29 Testing - Investigators | Rapid Onsite COVID-29 Testing - Participants | Total
Number analyzed (Participants) | 10 | 83 | 93
Age, Customized [Count of Participants; unit: Participants] — Population: Participant age was not collected.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Participant gender was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 83 | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Samples Tested
Description: samples are tested and consistently shown that the assay can detect SARS-CoV-2 safely, consistently and accurately at multiple locations using the mobile laboratory.
Time Frame: 15 minutes
Population: 3692 samples were collected from 93 participants.
Measure: Count of Units; unit: samples
Units Other Than Participants: samples
Arm/Group | Rapid Onsite COVID-29 Testing
Number analyzed (Participants) | 93
Number analyzed (samples) | 3692
samples | 3692

2. Primary Outcome: Safety: Number of Participants Who Tested Positive for COVID-19
Description: Feasibility is determined when at least 10000 samples are tested and consistently shown that the assay can detect SARS-CoV-2 safely, consistently and accurately at multiple locations using the mobile laboratory. This testing protocol will be considered safe if COVID-19 rates of those performing the tests do not significantly exceed those of the communities in which the tests are being performed.
Time Frame: up to 2 months
Population: The participants included people from the community and team members performing the tests.
Measure: Count of Participants; unit: Participants
Groups:
- Community Participants: Community participants that gave samples
- Investigator Participants: The team members that participated in the testing
Arm/Group | Community Participants | Investigator Participants
Number analyzed (Participants) | 83 | 10
Participants | 16 | 0

ADVERSE EVENTS:
Time Frame: Participants were not monitored for adverse events during sample collection.
Description: Participants were able to donate a saliva sample using two different methods. The first being a drop box with no interaction with the study team (saliva samples were collected off site) and the second being an in person saliva sample collection at designate dates and times. Participants were not monitored for adverse events during sample collection.
Groups:
- Rapid Onsite COVID-29 Testing - Community Participants: Community participants provide a saliva sample for a simple test to detect high concentrations of SARS-CoV-2 in saliva with assays that require no specialized equipment and can be completed in one hour.
  Rapid Onsite COVID-19 Detection: saliva assay test for high concentrations of SARS-CoV-2
- Rapid Onsite COVID-29 Testing - Investigator Participants: Investigator participants provide a saliva sample for a simple test to detect high concentrations of SARS-CoV-2 in saliva with assays that require no specialized equipment and can be completed in one hour.
  Rapid Onsite COVID-19 Detection: saliva assay test for high concentrations of SARS-CoV-2
Arm/Group | Rapid Onsite COVID-29 Testing - Community Participants | Rapid Onsite COVID-29 Testing - Investigator Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT04460690/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT04460690/ICF_000.pdf